CLINICAL TRIAL: NCT00082108
Title: National Registry of Myotonic Dystrophy and Facioscapulohumeral Muscular Dystrophy Patients and Family Members
Brief Title: Myotonic Dystrophy and Facioscapulohumeral Muscular Dystrophy Registry
Status: Recruiting | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Johanna Hamel, Associate Professor of Neurology, University of Rochester
Other Study IDs: NIAMS-104; U54NS048843 (NIH)
Record Dates: First submitted 2004-04-29; First posted 2004-04-30 (Estimated); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Myotonic Dystrophy; Facioscapulohumeral Muscular Dystrophy; Muscular Dystrophy; Myotonic Dystrophy Type 1; Myotonic Dystrophy Type 2; Congenital Myotonic Dystrophy; PROMM (Proximal Myotonic Myopathy); Steinert's Disease; Myotonic Muscular Dystrophy
Keywords: Registry; FSHD; DM; Muscular Dystrophy; Facioscapulohumeral Myotonic Dystrophy; Myotonic Dystrophy; DM1; DM2; FSH; MMD
MeSH Terms: conditions — Myotonic Dystrophy; Muscular Dystrophy, Facioscapulohumeral; Muscular Dystrophies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Myotonic dystrophy (DM) and facioscapulohumeral muscular dystrophy (FSHD) are inherited disorders characterized by progressive muscle weakness and loss of muscle tissue. The purpose of this registry is to connect people with DM or FSHD with researchers studying these diseases. The registry will offer individuals with DM and FSHD an opportunity to participate in research that focuses of their diseases. The registry will also help scientists to accomplish research on DM and FSHD and to distribute their findings to patients and care providers.

DETAILED DESCRIPTION:
The National Registry of DM and FSHD Patients and Family Members was developed to create a link between patients and scientists in order to promote research on these rare illnesses. The Registry is sponsored by the National Institutes of Health.

Patients that are interested in joining the Registry can email or call to request an application or download the forms from the website (www.dystrophyregistry.org). The Application packet contains:

* A Patient Information Form, which asks about your muscle strength, general health, and how your disease affects your daily life
* A Medical Records Release Form, which allows us to contact your doctor and obtain records about your diagnosis
* An informed Consent Form, which describes the study's purpose and what you can expect while you are involved with the project.

After you are enrolled in the Registry, there are several ways to participate in research. The activities include:

* Complete an annual update form to help us keep track of how your symptoms change over time.
* Receive updates about the progress of the Registry, research highlights, and other news related to muscular dystrophy through newsletters, an email listserv, and Facebook.
* Receive letters from the Registry when researchers are looking for patients to take part in studies. These projects may include filling out questionnaires, exploring new treatments, and other types of research.

There is no obligation to participate in these activities. Taking part in any study or filling out the annual updates are completely up to you.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with DM, FSHD, or related diseases or are an unaffected family member of someone diagnosed with one of these diseases

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will volunteer to participate in this study. The study will be advertised through neuromuscular disease clinics, the National Registry website, Patient Advocacy Groups and MDA Clinics through out the United States.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2000-09; Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Patient reported outcomes | Annual

CONTACTS AND LOCATIONS:
Overall Officials: Johann Hamel, MD, Principal Investigator — University of Rochester Medical Center, Department of Neurology
Locations (1):
- University of Rochester Medical Center, Department of Neurology, Rochester, New York, United States

REFERENCES:
- See also: Click here for more information about the National Registry. — http://www.dystrophyregistry.org
- See also: Click here for the National Registry's Facebook page. — https://www.facebook.com/NationalRegistryofMyotonicDystrophyandFSHD?ref=bookmarks